CLINICAL TRIAL: NCT05085119
Title: Validation of the Relationship Between Oxygenation Parameters and the Oxygen Reserve Index (ORI™), in Mechanically Ventilated ICU Patients: An Exploratory Pathophysiology Study
Brief Title: Validation of the Relationship Between Oxygenation Parameters and ORI™, in Mechanically Ventilated ICU Patients
Acronym: FiO2RI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RBHP 2019 GODET 3
Record Dates: First submitted 2021-09-15; First posted 2021-10-20 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Intubation; Mechanical Ventilation; Intensive Care Unit
Keywords: Oxygen administration; Oxygen blood content; ORI; Intensive care unit; ICU; Mechanical ventilation; Intubation

STUDY DESIGN:
Intervention Model Description: Validation study of a non-invasive sensor-type medical device, with comparison to standard paraclinical parameters, with a stepwise modification test of FIO2, in normo- to moderate hyperoxic conditions.
Masking Description: FiO2 steps will be conducted by study investigator. Participants, care providers and outcomes assessor will remain blinded of FiO2 steps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FiO2 stepwise modifications (Experimental): Intubation ICU patients will be challenged with stepwise modifications of FiO2. The following steps will be done: 30, 40, 60, 80, 100, 80, 60, 40 and 30%.
  Interventions: Procedure: Stepwise modifications of FiO2

INTERVENTIONS:
Procedure: Stepwise modifications of FiO2 — FiO2 will be increased stepwise from 30 to 100% (40, 60 and 80%), and then decreased with the same FiO2 reverse steps.

SUMMARY:
The ORI™ or Oxygen Reserve Index (Masimo, Irvine, CA, USA) is a non-invasive monitoring system for measuring oxygen reserve. It is a digital sensor (almost identical to the SpO2 sensor) which allows an analysis of the absorption of arterial, venous and capillary components. The measured index, unitless, ranges from 0.00 to 1.00 for moderate hyperoxia levels: from 100 to 200 mmHg. It can alert the clinician to a drop in oxygen stores via the drop in SvO2 before a drop in SpO2 is observed. We propose to carry out a study to elucidate correlation between ORI™ and PaO2.

DETAILED DESCRIPTION:
Pulse oximetry or SpO2 is the standard and mandatory monitoring of oxygenation during mechanical ventilation of intensive care and operating theatre patients. Its use is based on the difference in infrared and red light absorptions of oxyhaemoglobin and reduced haemoglobin. The calculation of the absorption percentage takes into account the pulsatility of the signal, reflecting the arterial component, while eliminating the continuous signal, reflecting the venous component. It is then considered that SpO2 is a reflection of SaO2, or arterial oxygen saturation. Oxygen exists in two forms in the arterial circulation: dissolved (PaO2) or bound to haemoglobin (SaO2).

Because of the sigmoidal shape of the oxyhaemoglobin dissociation curve, SpO2 is a late marker of arterial hypoxaemia. Indeed, SpO2 only starts to decrease after a marked drop in PaO2.

Hypoxaemia is a frequent situation, both in the operating theatre during the period of securing the airway, intra-operatively, or post-operatively, after extubation, on episodes of alveolar hypoventilation, such as atelectasis. In intensive care units, it can occur in injured lungs with various aetiologies (infectious, inflammatory, cardiac, etc). It is an independent predictive factor of mortality.

Exposure of patients to high hyperoxia (FiO2>0.7), over a long period of time, can lead to pulmonary endothelial damage (due to the formation of reactive oxygen species, ROS), denitrogenation atelectasis, and possibly a systemic inflammatory cascade. It is currently suggested that hyperoxia may also have a haemodynamic impact, with a fall in cardiac output and peripheral vasoconstriction, particularly in healthy volunteers and patients with cardiac decompensation. However, hyperoxia is a frequent situation during the perioperative period as it provides safety and a potential oxygen reserve in case of adverse events: hemodynamic degradation, cardiac arrest, extubation...

The ORI™ or Oxygen Reserve Index (Masimo, Irvine, CA, USA) is a non-invasive monitoring system for measuring oxygen reserve. It is a digital sensor (almost identical to the SpO2 sensor) which allows an analysis of the absorption of arterial, venous and capillary components. The measured index, unitless, ranges from 0.00 to 1.00 for moderate hyperoxia levels: from 100 to 200 mmHg. It can alert the clinician to a drop in oxygen stores via the drop in SvO2 before a drop in SpO2 is observed.

There is little literature on ORI™. A previous study showed a poor correlation between ORI™ (ranging from 0.24 to 0.55) and PaO2, which ranged from 100 to 150 mmHg, respectively. The company, Masimo, has recently made a change in its algorithm, allowing it to re-calibrate its sensor. However, no new correlation research has been conducted. We therefore propose to carry out a new test phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years, admitted in an intensive care unit of the Peri-Operative Medicine Pole of the Clermont-Ferrand University Hospital, under invasive mechanical ventilation (intubation or tracheotomy), whose FiO2 required to obtain an SpO2 > 95% is ≤ 30%, equipped as part of routine care with an arterial catheter and a central venous catheter in the superior vena cava territory
* BMI < 30 kg.m-2
* Written consent to participate in the study by the patient or by the trusted person, or the relative if he or she is present.

Exclusion Criteria:

* Existence of an underlying pulmonary pathology that may alter oxygen diffusion or generate an intra-pulmonary shunt (COPD, emphysema, pneumopathy, ARDS, chronic respiratory failure...)
* Uncontrolled haemodynamic instability defined by an increase of more than 20% in catecholamine dosages during the last hour, despite optimisation of the blood volume according to a pre-established protocol (mini-fluid challenge)
* Patient already included in the study
* Patient's or relative's refusal to participate
* Guardianship or trusteeship patient
* No affiliation to the Social Security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Correlation between ORI™ and PaO2 | There will be nine 10 minutes steps. Measurement will be done during the last minute of each 10 minutes step
  Correlations will be investigated during the last minute of each 10 minutes FiO2 steps

SECONDARY OUTCOMES:
Correlation between ORI™ and PcvO2 | There will be nine 10 minutes steps. Measurement will be done during the last minute of each 10 minutes step
  Correlations will be investigated during the last minute of each 10 minutes FiO2 steps
Correlation between ORI™ and ScvO2 | There will be nine 10 minutes steps. Measurement will be done during the last minute of each 10 minutes step
  Correlations will be investigated during the last minute of each 10 minutes FiO2 steps
Correlation between ORI™ and SaO2 | There will be nine 10 minutes steps. Measurement will be done during the last minute of each 10 minutes step
  Correlations will be investigated during the last minute of each 10 minutes FiO2 steps
Correlation between ORI™ and SpO2 | There will be nine 10 minutes steps. Measurement will be done during the last minute of each 10 minutes step
  Correlations will be investigated during the last minute of each 10 minutes FiO2 steps

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - CHU, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: Undecided